CLINICAL TRIAL: NCT02388620
Title: A Phase I, Open Label, Multi-center, Parallel Cohort, Single Dose Study to Evaluate the Pharmacokinetics of LEE011 in Healthy Subjects With Normal Hepatic Function and Subjects With Impaired Hepatic Function.
Brief Title: Evaluation of Hepatic Function Impairment on the Pharmacokinetics of LEE011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A2109
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-12

CONDITIONS: Normal Hepatic Function; Impaired Hepatic Function
MeSH Terms: interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Experimental): Normal hepatic function; matched demography to hepatic impairment cohorts
  Interventions: Drug: LEE011
- Mild Hepatic Impairment (Experimental): Child-Pugh Classification A (score 5-6)
  Interventions: Drug: LEE011
- Moderate Hepatic Impairment (Experimental): Child-Pugh Classification B (score 7-9)
  Interventions: Drug: LEE011
- Severe Hepatic Impairment (Experimental): Child-Pugh Classification C (score 10-15)
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011 — 400 mg
  Other Names: Ribociclib

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety and tolerability of a single oral dose of LEE011 in subjects with varying degrees of impaired hepatic function (based on Child-Pugh classification) as compared to demographically-matched control subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

Male or female (sterile or postmenopausal) subjects between 18-75 (both inclusive) years of age and healthy as determined by absence of clinically significant deviation from normal in medical history, physical examination, vital signs, electrocardiograms, and clinical laboratory determinations.

Subjects must have a BMI between 18 kg/m2 and 36 kg/m2 and weight at least 50 kg and no more than 120 kg.

Other than hepatic impairment, subjects must be in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, (except for additional inclusion criteria described below).

Subjects in Child-Pugh A, B and C cohorts: Additional inclusion criteria

Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment

No change in hepatic status at least one month prior to dosing (i.e. worsening of Child-Pugh score).

Exclusion Criteria:

All Subjects:

Subject has received a liver transplant at any time in the past and is on immunosuppressant therapy.

History or presence of impaired cardiac function

Any surgical or medical condition that may significantly alter the absorption, distribution, metabolism or excretion of drugs

Administration of CYP3A4/5 inhibitors or inducers or CYP3A4 substrates with narrow therapeutic windows

Administration of medications that prolong the QT interval

History of immunodeficiency diseases, including HIV, as confirmed by (HIV-1, HIV-2) test.

Participation in another clinical trial within 4 weeks prior to the study drug administration.

Subjects with normal hepatic function:

Additional exclusion criteria A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Subjects in Child-Pugh A, B and C cohorts:

Additional exclusion criteria

Clinical evidence of severe ascites (e.g. requiring regular tapping).

Bilirubin > 6 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Composite Pharmacokinetic (PK) profile of a single oral dose of LEE011 in subjects with impaired hepatic function as compared to healthy subjects with normal hepatic function. | 14 days
  PK profile includes the following parameters Tmax, Cmax, AUClast, AUCinf, T1/2, CL/F, Vz/F.

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) | From consent to 28 days post-dose
  Safety profile of a single dose of LEE011 in healthy subjects and subjects with varying degrees of hepatic function includes changes observed in physical examination, changes in vital signs, changes in electrocardiograms (ECGs), abnormal laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - University of Miami, Coral Gables, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samant TS, Yang S, Miller M, Ji Y. Pharmacokinetics of Ribociclib in Subjects With Hepatic Impairment. J Clin Pharmacol. 2021 Aug;61(8):1001-1009. doi: 10.1002/jcph.1825. Epub 2021 Mar 12. PMID 33555033
- See also: Results for CLEE011A2109 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16928